CLINICAL TRIAL: NCT04907422
Title: Gold Nanoparticles as Novel Biomarkers for Cancer Stem Cells in Salivary Gland Tumors: A Diagnostic and Prognostic Accuracy Study
Brief Title: Diagnostic and Prognostic Accuracy of Gold Nanoparticles in Salivary Gland Tumours
Status: Completed | Type: Observational
Sponsor: Amina Fouad Farag (Other)
Responsible Party: Sponsor-Investigator, Amina Fouad Farag, Lecturer of Oral and Maxillofacial Pathology, Oral Pathology Department, Faculty of Dentistry, October 6 University
Organization: October 6 University (Other)
Other Study IDs: RECO6U/5-2018
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma Ex Pleomorphic Adenoma of Salivary Glands; Pleomorphic Adenoma of Salivary Glands
Keywords: Cancer stem cells; CD24-Gold Nanocomposite; CD24; Gold nanoparticles; Sensitivity; Specificity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Briefly, a portion of surgically resected salivary gland tumour specimens was immersed immediately in liquid nitrogen, allowed to snap frozen and stored at -80 C (Frozen tissue) while the other portion was fixed in 10% buffered formalin solution and embedded in paraffin (Formalin-fixed paraffin-embedded tissue)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CXPA group: carcinoma ex pleomorphic adenoma of major and minor salivary glands.
  Interventions: Diagnostic Test: CD24-Gold Nanocomposite expression using Real-time quantitative polymerase chain reaction; Diagnostic Test: non-conjugated CD24 expression using Real-time quantitative polymerase chain reaction
- PA group: Benign pleomorphic adenoma of major and minor salivary glands.
  Interventions: Diagnostic Test: CD24-Gold Nanocomposite expression using Real-time quantitative polymerase chain reaction; Diagnostic Test: non-conjugated CD24 expression using Real-time quantitative polymerase chain reaction
- Control group: normal controls obtained from border of excision biopsy of mucocele in the lip mucosa of healthy individuals.
  Interventions: Diagnostic Test: CD24-Gold Nanocomposite expression using Real-time quantitative polymerase chain reaction; Diagnostic Test: non-conjugated CD24 expression using Real-time quantitative polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: CD24-Gold Nanocomposite expression using Real-time quantitative polymerase chain reaction — new strategy where gold nanoparticles synthetized and added to CD24 primer forming CD24-Gold Nanocomposite to be used for detection of cancer stem cells
  Other Names: CD24-AuNC expression using Real-time qPCR
Diagnostic Test: non-conjugated CD24 expression using Real-time quantitative polymerase chain reaction — conventional strategy using non-conjugated CD24 expression to used for detection of cancer stem cells
  Other Names: CD24 expression using Real-time qPCR

SUMMARY:
Nano-based diagnostic tool can provide promising highly sensitive, specific biomarker for early detection and treatment of salivary gland tumours compared to non-conjugated biomarkers and in turn improves patient prognosis and outcome.

DETAILED DESCRIPTION:
Cancer stem cells form a small subset of highly tumorigenic cells within the bulk of the tumours which mainly responsible for initiation, invasion, rapid growth, metastasis and therapeutic resistance in different types of human cancers. Nowadays, nanotechnology has increasing attention in multi-disciplinary research fields. Conjugated gold nanoparticles are widely used as biomarkers and bio-delivery vehicles in the medicine as well as early and advanced cancer detection and treatment. The current work aimed to introduce a novel diagnostic and prognostic approach in early detection of cancer stem cells in salivary gland tumours using gold nanoparticles conjugated to CD24 (CD24-Gold Nanocomposite).

ELIGIBILITY:
Inclusion Criteria:

* Benign PA of major and minor salivary glands (PA group),
* CXPA of major and minor salivary glands (CXPA group).
* Border of excision biopsy of mucocele in the lip mucosa of healthy individuals used as normal controls (Control group).
* Surgical excision of tumors with no preoperative chemotherapy or radiotherapy. For parotid tumours partial or total parotidectomy, Surgery was performed with or without facial nerve preservation and the later was carried out commonly when the nerve was involved by tumour. For tumours in the other glands, complete surgical excision with the involved gland and the suspicious adjacent structures was performed.

Exclusion Criteria:

* All epithelial origin salivary gland tumours other than PA and CXPA.
* All mesenchymal origin salivary gland tumours.
* All inflammatory and cystic lesions of salivary glands.
* Metastasis in salivary glands.
* Patients received preoperative chemotherapy or radiotherapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presented to Oral and Maxillofacial Surgery Department, Faculty of Dentistry and Output Clinics of General Surgery Department, Faculty of Medicine, October 6 University, Giza, Egypt.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic potential of CD24-AuNC (index test) compared to non-conjugated CD24 (reference test) in determination of salivary gland tumours | Done immediately following completion of assessment for eligibility of enrolment in the present study (enrolment took about 6 months) and confirmation of definite diagnosis
  we tested the differential expression of CD24-AuNC and non-conjugated CD24 biomarkers in all studied groups in order to identify the most sensitive and specific diagnostic biomarker to be used in detecting salivary gland tumours,

SECONDARY OUTCOMES:
Clinicopathological characteristics of the patients and their association with CD24-AuNC (Index test) and non-conjugated CD24 (Reference test) expressions | Done immediately following completion of assessment for eligibility of enrolment in the present study (enrolment took about 6 months) and confirmation of definite diagnosis
  We investigated the relationship between both biomarkers' expression and clinicopathological characteristics of PA and CXPA patients such as age, gender, tumor site, tumor size (maximum diameter in mm), histopathological subtype, encapsulation, degree of invasion, facial nerve involvement and lymph node (LN) metastasis that may have direct relation with the tumor prognosis
Prognostic significance of CD24-AuNC (index test) compared to non-conjugated CD24 (reference test) in assessing disease progression and/or patient survival | At regular intervals every 3 months for 24-months (follow-up period)
  we assessed the disease progression and/or patient survival and examined its association with biomarkers expression

CONTACTS AND LOCATIONS:
Overall Officials: Amina F Farag, PhD, Principal Investigator — Faculty of Dentistry, October 6 University
Locations (1):
- Faculty of Dentistry, October 6 University, Giza, Egypt

REFERENCES:
- [Derived] Kesharwani P, Ma R, Sang L, Fatima M, Sheikh A, Abourehab MAS, Gupta N, Chen ZS, Zhou Y. Gold nanoparticles and gold nanorods in the landscape of cancer therapy. Mol Cancer. 2023 Jun 21;22(1):98. doi: 10.1186/s12943-023-01798-8. PMID 37344887
- [Derived] Farag AF, Hassabou NF. CD24-gold nanocomposite as promising and sensitive biomarker for cancer stem cells in salivary gland tumors. Nanomedicine. 2022 Nov;46:102598. doi: 10.1016/j.nano.2022.102598. Epub 2022 Sep 8. PMID 36089234